CLINICAL TRIAL: NCT03679806
Title: Effects Aquatic Exercises on Balance and Hand Function in Multiple Sclerosis: Halliwick Versus Aquatic Plyometric Exercises
Brief Title: Effects Aquatic Exercises on Balance and Hand Function in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Barış Gürpınar, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: msdexerity
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: aquatic therapy; Limits of stability; Halliwick; aquatic plyometric exercises
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Halliwick (Experimental): Exercises were performed in a private pool owned by the local MS society twice in a week for 8 weeks. Pool depth was 120 cm 30-31°C Mental adjustment, sagittal rotation, transverse rotation, and combined rotation controls, balances in stillness steps of the Halliwick concept were included.
  Interventions: Other: Halliwick
- Aquatic Plyometric Exercise (Experimental): Exercises were performed in a private pool owned by the local MS society twice in a week for 8 weeks. Pool depth was 120 cm 30-31°C. The three phases of each exercise; eccentric (or loading) phase, the amortization phase, and the concentric (or unloading) phase included.
  Interventions: Other: Aquatic Plyometric Exercises

INTERVENTIONS:
Other: Halliwick — The exercise program was progressed by increasing the speed and the range of motion of the movements. Patients were asked not to accelerate the exercise and to focus on their alignment. Mental adjustment, sagittal rotation, transverse rotation, and combined rotation controls, balances in stillness steps of the Halliwick concept were included.
  Arms: Halliwick
Other: Aquatic Plyometric Exercises — The APE programme was progressed by increasing speed and the range of motion of the movements. Patients were carefully informed not to deform the exercise just to emulate the speed. The three phases of each exercise; eccentric (or loading) phase, the amortization phase, and the concentric (or unloading) phase explained thoroughly at the beginning of every exercise.
  Arms: Aquatic Plyometric Exercise

SUMMARY:
This study aims to compare and contrast the effects of two different aquatic exercises on postural control and hand functions in people with multiple sclerosis.

DETAILED DESCRIPTION:
Impaired limits of stability causes falls in people with Multiple sclerosis (pwMS) whereas a well-controlled posture provides improved upper limb functions which are limited in almost 75% of pwMS due to weakness, spasticity or tremor. It is an already known fact that hand dexterity is an indicator of fall risk due to neuromuscular causes and/or abnormalities in the corpus callosum in pwMS.

Aquatic therapy (AT) provides a safe and effective environment for many therapeutic purposes. It is important to understand the effects of each type, intensity, and duration of the aquatic interventions to accomplish most suitable aquatic exercise program.

Halliwick method, neuromotor treatment approach which uses fluid and mechanical properties of water, is based on postural control by mobilizing and controlling body parts through the Ten Point Program.

During Aquatic Plyometric Exercises, proximal part of the body needs to be stabilized to generate a sudden and powerful contraction at the distal part and stabilization of the proximal joints is necessary for maintaining distal movements in a coordinated way.

It is important to understand the effects of each type, intensity, and duration of the aquatic interventions to accomplish most suitable aquatic exercise program. This study aims to compare and contrast the effects of two different aquatic exercises on postural control and hand function.

ELIGIBILITY:
Inclusion Criteria:

* EDSS>6
* volunteered

Exclusion Criteria:

* Clinical relapse within three months
* incontinence
* persistent infection

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in limits of stability | Baseline and 8 weeks
  measured with Biodex Balance System (BBS; SD 12.1"Display 115 VAC). Patients were asked to stand on the rigid surface with barefoot and eyes open during measuring limits of stability. During each test trial, patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. The same process is repeated for each of the nine targets. Targets on the screen blink in random order. The tests repeated three times with 30 second resting time between trials. Patients' performance is evaluated from a total score of 100 where the higher score represents better trunk control.
Change in Nine hole peg Test | Baseline and 8 weeks
  The patient is seated at a table with a plastic NHPT placed at the patient's middle and asked to place pegs in a random order as quick as possible by using dominant hand first total time was recorded in seconds. Three consecutive trials with the dominant hand are immediately followed by three consecutive trials with the non-dominant hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No